CLINICAL TRIAL: NCT06530498
Title: Diagnostics of Clinical Hyperandrogenism Using the Modified Ferriman-Gallwey Scale and the Ludwig Scale in Women With Normogonadotropic Anovulation
Brief Title: Diagnostics of Clinical Hyperandrogenism
Status: Recruiting | Type: Observational
Sponsor: Jagiellonian University (Other)
Responsible Party: Principal Investigator, Iwona Magdalena Gawron, MD, PhD, Jagiellonian University
Other Study IDs: 118.0043.1.24.2024
Record Dates: First submitted 2024-07-28; First posted 2024-07-31 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Anovulation; PCOS
Keywords: Hirsutism; Normogonadotropic Anovulation; PCOS; androgenetic alopecia
MeSH Terms: conditions — Anovulation; Hirsutism; Alopecia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Polycystic ovary syndrome (PCOS): Women diagnosed with polycystic ovary syndrome based on International Evidence-based Guideline for the assessment and management of polycystic ovary syndrome (2023)
  Interventions: Diagnostic Test: Assessment of the severity of hirsutism using the visual modified Ferriman-Gallwey scale; Diagnostic Test: Assessment of the severity of endogenetic alopecia using the visual Ludwig Scale
- Hypothalamic-pituitary-ovarian dysfunction (HPOD): Women diagnosed with hypothalamic-pituitary-ovarian dysfunction based on The FIGO ovulatory disorders classification system (2022)
  Interventions: Diagnostic Test: Assessment of the severity of hirsutism using the visual modified Ferriman-Gallwey scale; Diagnostic Test: Assessment of the severity of endogenetic alopecia using the visual Ludwig Scale

INTERVENTIONS:
Diagnostic Test: Assessment of the severity of hirsutism using the visual modified Ferriman-Gallwey scale — Assessment of the severity of hirsutism using the visual modified Ferriman-Gallwey scale in 9 body regions rated from 0 (no growth of terminal hair) to 4 (extensive hair growth), thus with a score ranging from 0 (the lowest score - no hirsutism) to 36 points (the highest score - the greatest severity of hirsutism)
Diagnostic Test: Assessment of the severity of endogenetic alopecia using the visual Ludwig Scale — Visual assessment of baldness on the Ludwig scale from I (least severe baldness) to III (most severe baldness):
  Type I - minimal thinning of the mid-line parting in the hair; Type II - gradual thinning and noticeable widening of the mid-line parting in the hair; Type III - Heavy to total thinning of the mid-line

SUMMARY:
The optimal cut-off value for diagnosing hirsutism in the modified Ferriman-Gallwey (mFG) point scale in the Polish population is not known. The correlation of mFG with the severity of androgenetic alopecia in the Ludwig scale (LS) is not known.

The aim of the study is to determine the cut-off point for the diagnosis of hirsutism and to assess the correlation of the mFG scale score with the LS of androgenetic alopecia severity.

DETAILED DESCRIPTION:
The aim of the study is to:

* determine the cut-off point on the mFG scale, indicating hirsutism and to determine the correlation of the severity of androgenetic alopecia on the Ludwig scale with the mFG value in the population of women diagnosed and treated at the University Hospital in Krakow due to anovulation.
* to determine the severity of hirsutism and the severity of androgenetic alopecia in individual PCOS phenotypes.

Inclusion criteria are as follows: i) oligoovulation, i.e. menstrual cycles every <21 days or >35 days, ii) age 18-45 years, iii) diagnosis of PCOS.

Exclusion criteria: none.

To achieve the study objectives, the following will be performed:

* Visual assessment of the severity of hirsutism on the modified Ferriman-Gallwey scale
* Visual assessment of the severity of androgenetic alopecia on the Ludwig scale.

ELIGIBILITY:
Inclusion Criteria:

* oligoovulation, i.e. menstrual cycles every <21 days or >35 days
* age 18-45 years
* diagnosis of PCOS.

Exclusion Criteria:

* none

Ages: 18 Years to 45 Years | Sex: Female
Age Groups: Adult
Study Population: Women diagnosed and treated at the University Hospital in Krakow due to normogonadotropic anovulation
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-02-08 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Comparison of the severity of hirsutism in the PCOS and HPOD groups | up to 6 months
  Comparison of the mFG score in the PCOS and HPOD groups; The modified Ferriman-Gallwey (mFG) scale assesses the severity of excessive hair growth on a scale of 0-4 points in 9 body regions (Upper lip, Chin, Chest, Upper back, Lower back, Upper abdomen, Lower abdomen, Upper arms, Thighs); the lowest possible score is 0 and the highest is 36; the higher the score, the greater the severity of excess hair
Comparison of the severity of endogenetic alopecia in the PCOS and HPOD groups | up to 6 months
  Comparison of the LS score in the PCOS and HPOD groups; The Ludwig Scale (LS) assesses the severity of androgenetic alopecia on a scale from I to III, with additional sub-points within some of the above grades, i.e. I-1, I-2, I-3, I-4, II-1, II-2, III, IV (frontal - advanced); the higher the grade, the greater the severity of alopecia
Calculation of cut-off point for diagnosing hirsutism in the study population | up to 6 months
  The cut-off point for diagnosing hirsutism will be calculated using the receiver operating characteristic curve
Assessment of diagnostic convergence of mFG and LS scales in diagnosing clinical hyperandrogenism | up to 6 months
  The correlation of mFG and LS scale scores in the study population will be assessed using standard statistical methods

CONTACTS AND LOCATIONS:
Overall Officials: Kazimierz Pityński, Prof., PhD, MD, Study Chair — Jagiellonian University
Locations (1):
- Jagiellonian University Medical College, Krakow, Poland